CLINICAL TRIAL: NCT04556786
Title: The Impact of a Pharmacist-Led Transitional Care Program on Health Outcomes of Uninsured Populations
Brief Title: A Pharmacist-led Transitions of Care Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Chiahung Chou, Ph.D., Associate Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-342 EX 1809
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Chronic Disease
Keywords: Transitions of care; Indigent population; Hospital readmission rates
MeSH Terms: conditions — Chronic Disease | interventions — Patient Transfer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitions of care (Experimental): The study participants in this aim received usual care plus medication reconciliation, daily schedule for medication taking and medical condition monitoring, and follow-up phone calls from a pharmacist.
  Interventions: Behavioral: Transitions of care
- Usual care (No Intervention): The study participants in this arm received usual care.

INTERVENTIONS:
Behavioral: Transitions of care — The intervention was a pharmacist-led transitions of care program that include medication reconciliation, daily schedule for medication taking and medical condition monitoring, and follow-up phone calls from a pharmacist at 60- and 90-day post-discharge in addition to the usual care.
  Arms: Transitions of care

SUMMARY:
This study was to show the value of pharmacists in providing transitions of care to and improving health outcomes of uninsured populations. It also aimed to demonstrate the feasibility of implementing a transitions of care program in an indigent care clinic with limited resources. We hypothesized that a pharmacist-led transitions of care program will reduce 30-day hospital readmission rates among the uninsured discharged from a community hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older
* Uninsured
* English speaking
* Discharged from East Alabama Medical Center within the past 16 days

Exclusion Criteria:

* Patients who did not show up for the first follow-up visit with the study pharmacist after being referred by the care coordinator at East Alabama Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
30-day hospital readmission | 30-day post-discharge
  Whether a study participant had any hospital readmission 30-day post-discharge

SECONDARY OUTCOMES:
60-day hospital readmission | 60-day post-discharge
  Whether a study participant had any hospital readmission 60-day post-discharge
90-day hospital readmission | 90-day post-discharge
  Whether a study participant had any hospital readmission 90-day post-discharge
30-day emergency department (ED) visit | 30-day post-discharge
  Number of ED visits among study participants in each study arm 30-day post-discharge
60-day emergency department (ED) visit | 60-day post-discharge
  Number of ED visits among study participants in each study arm 60-day post-discharge
90-day emergency department (ED) visit | 90-day post-discharge
  Number of ED visits among study participants in each study arm 90-day post-discharge
30-day follow-up visit with a primary care provider | 30-day post-discharge
  Did a study participant keep a follow-up appointment with a primary care provider

CONTACTS AND LOCATIONS:
Overall Officials: Chiahung Chou, PhD, Principal Investigator — Auburn University
Locations (1):
- Mercy Medical Clinic, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Englander H, Kansagara D. Planning and designing the care transitions innovation (C-Train) for uninsured and Medicaid patients. J Hosp Med. 2012 Sep;7(7):524-9. doi: 10.1002/jhm.1926. Epub 2012 Mar 12. PMID 22411913
- [Background] Hawes EM, Maxwell WD, White SF, Mangun J, Lin FC. Impact of an outpatient pharmacist intervention on medication discrepancies and health care resource utilization in posthospitalization care transitions. J Prim Care Community Health. 2014 Jan 1;5(1):14-8. doi: 10.1177/2150131913502489. Epub 2013 Sep 17. PMID 24327590
- [Background] Crotty M, Rowett D, Spurling L, Giles LC, Phillips PA. Does the addition of a pharmacist transition coordinator improve evidence-based medication management and health outcomes in older adults moving from the hospital to a long-term care facility? Results of a randomized, controlled trial. Am J Geriatr Pharmacother. 2004 Dec;2(4):257-64. doi: 10.1016/j.amjopharm.2005.01.001. PMID 15903284
- [Background] Phatak A, Prusi R, Ward B, Hansen LO, Williams MV, Vetter E, Chapman N, Postelnick M. Impact of pharmacist involvement in the transitional care of high-risk patients through medication reconciliation, medication education, and postdischarge call-backs (IPITCH Study). J Hosp Med. 2016 Jan;11(1):39-44. doi: 10.1002/jhm.2493. Epub 2015 Oct 5. PMID 26434752
- See also: Key Facts about the Uninsured Population — http://files.kff.org/attachment/Fact-Sheet-Key-Facts-about-the-Uninsured-Population
- See also: America's Health Rankings — https://assets.americashealthrankings.org/app/uploads/ahrannual17_complete-121817.pdf